CLINICAL TRIAL: NCT01825486
Title: Balance and Gait Characteristics to Predict Accidental Falls in Community-dwelling Stroke Elderly
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Other Study IDs: I050309
Record Dates: First submitted 2013-04-03; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Cerebrovascular Accident; Accidental Falls
Keywords: Balance; Gait characteristics
MeSH Terms: conditions — Stroke | interventions — Accidental Falls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- accidental falls
  Interventions: Behavioral: accidental falls

INTERVENTIONS:
Behavioral: accidental falls

SUMMARY:
Background: Accidental falls result in major physical and psychological morbidity in the elderly, especially stroke patients. To get optimal prevention of stroke falls, it is crucial to identify independent risk factors from multivariate analysis of related balance and gait parameters.

Aim: To evaluate the effects of balance and gait characteristics in determining whether or not accidental falls may happen. To investigate if the balance and gait parameters affect the time from lesion to when (and if) patients suffer from falls. To compare differences of balance and gait parameters in accidental fall patients between those with severe accidental injuries and those without severe injuries.

Methods: The 2-year observational cohort study will enroll 706 elderly stroke patients, who have not had a previous stroke. They will be retrieved from the Inpatient department and followed-up regularly in the Outpatient department when they are discharged. All subjects will be evaluated at 1 month and 6 months after stroke. These evaluations will include: mental, cognition and depression status; lower-limb muscle strength assessed by a dynamometer as well as range of motion of joints assessed by a biaxial electro-goniometry; functional independence measure; balance and gait pattern will be assessed by both clinical observation and objective laboratory examination (a dynamic posturography and computerized gait analysis system); falls and fall-related injuries during the proceeding year. Differences in baseline characteristics are tested by one-way ANOVA, Mann Whitney U or t tests, if appropriate. The investigators will identify the independent risk factors of accidental falls with logistic regression and use the log rank statistic of Kaplan-Meier survival curve to differentiate the risk of accidental falls or fall-related injuries in different groups.

ELIGIBILITY:
Inclusion Criteria:

* age>65
* confirmed stroke by CT or MRI
* first-ever stroke
* with walking ability after stroke onset 1 month

Exclusion Criteria:

* fall history before stroke
* living in nursing home
* unstable physical sign
* seizure attack during study
* impaired cognition

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: first-ever stroke patients were retrieved from the Inpatient department and followed-up regularly in the Outpatient department when they are discharged
Sampling Method: Non-Probability Sample
Dates: Start 2005-08; Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Computerized balance evaluation | 1 month after the first stroke
  computerized balance and gait evaluation by a posturography and gait analysis system

SECONDARY OUTCOMES:
Geriatric Depression Scale | 1 month after the first stroke
  Geriatric Depression Scale to measure depression

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital Taiwan, Changhua, Taiwan